CLINICAL TRIAL: NCT00553462
Title: A Phase II Study of Induction Chemotherapy Followed by Thoracic Radiotherapy and Erlotinib in Poor-Risk Stage III Non-Small Cell Lung Cancer
Brief Title: Carboplatin and Paclitaxel Albumin-Stabilized Nanoparticle Formulation Followed by Radiation Therapy and Erlotinib in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30605; CALGB-30605; CDR0000573832 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Erlotinib Hydrochloride; Taxes; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel + carboplatin + radiation + erlotinib (Experimental): Patients receive paclitaxel IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patient with rapid disease progression outside of the chest after induction therapy are removed from study.
  Patients with intrathoracic disease progression within the potential radiation field may continue protocol therapy at the discretion of the Study Chair. Patients with no disease progression outside the planned radiation field (either regional or distant) proceed to concurrent erlotinib hydrochloride and radiotherapy.
  Beginning on day 43 (week 7), patients receive oral erlotinib hydrochloride once daily. Patients also undergo concurrent radiotherapy 5 days a week for up to 7 weeks (33 fractions) in the absence of rapid disease progression outside of the chest or unacceptable toxicity.
  After completion of study therapy, patients are followed every 3 months for 1 year, and then every 6 months for up to 2 years
  Interventions: Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: erlotinib hydrochloride
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Erlotinib may make tumor cells more sensitive to radiation therapy. Giving carboplatin and paclitaxel albumin-stabilized nanoparticle formulation together with radiation therapy and erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and paclitaxel albumin-stabilized nanoparticle formulation together with radiation therapy and erlotinib works in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the activity of induction chemotherapy comprising carboplatin and paclitaxel albumin-stabilized nanoparticle formulation followed by concurrent thoracic radiotherapy and erlotinib hydrochloride in patients with poor-risk, unresectable stage IIIA or IIIB non-small cell lung cancer.

Secondary

* To determine the response rate and progression-free survival of these patients.

OUTLINE: Patients receive induction chemotherapy comprising paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patient with rapid disease progression outside of the chest after induction therapy are removed from study. Patients with intrathoracic disease progression within the potential radiation field may continue protocol therapy at the discretion of the Study Chair. Patients with no disease progression outside the planned radiation field (either regional or distant) proceed to concurrent erlotinib hydrochloride and radiotherapy.

Beginning on day 43 (week 7), patients receive oral erlotinib hydrochloride once daily. Patients also undergo concurrent radiotherapy 5 days a week for up to 7 weeks (33 fractions) in the absence of rapid disease progression outside of the chest or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 1 year, and then every 6 months for up to 2 years

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including any of the following histologies:

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar cell)
  * Large cell anaplastic carcinoma (including giant and clear cell carcinomas)
* Must meet the following criteria:

  * T1-3 with N2 and selected N3*
  * T4 with N0, N1, N2 and selected N3*
  * M0 (no M1 patients) NOTE: *Patients with contralateral mediastinal disease (i.e., N3) are eligible, provided all gross disease can be encompassed within the radiation boost field in accordance with the homogeneity criteria. Patients with ipsilateral scalene or supraclavicular disease are also eligible. Patients with contralateral hilar or supraclavicular node involvement are not eligible.
* Must have measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * Nonmeasurable lesions include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area
* Patients must be considered unresectable or inoperable AND be deemed candidates for combined modality therapy by a medical oncologist and a radiation oncologist
* Considered to be poor-risk with NCI CTC performance status (PS) 2 OR PS 0-1 and ≥ 10% weight loss within the past 3 months
* Patients with tumors adjacent to a vertebral body are eligible, provided all gross disease can be encompassed within the radiation boost field in accordance with the homogeneity criteria
* Pleural effusions meeting the following criteria allowed:

  * Effusion is transudate, cytologically negative, and non-bloody
  * Effusion can be seen on the chest CT scan but not on the chest x-ray AND is too small to tap
  * Effusion appears only after a thoracotomy or other invasive thoracic procedure was attempted

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Granulocytes ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* AST < 2 x ULN
* Bilirubin ≤ ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for NSCLC
* At least 2 weeks since formal exploratory thoracotomy
* No concurrent administration of sucralfate suspension and erlotinib hydrochloride
* No concurrent intensity-modulated radiotherapy
* No concurrent hormones or other chemotherapeutic agents except steroids given for adrenal failure, hormones administered for non-disease-related conditions (e.g., insulin for diabetes), and intermittent use of dexamethasone as an antiemetic
* No concurrent palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-03; Primary Completion 2014-01 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, MD, Study Chair — Cleveland Clinic Florida
Locations (99):
- United States (99):
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and October 2011, 78 participants were recruited to this study.
Pre-assignment Details: Three participants did not receive any protocol treatment and were excluded from all analyses.
Groups:
- Paclitaxel + Carboplatin + Radiation + Erlotinib: Patients receive paclitaxel 100 mg/m^2 IV over 30 minutes on days 1 and 8 and carboplatin AUC=5 IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses.
  Beginning on day 43 (week 7), patients receive oral erlotinib hydrochloride 150 mg once daily. Patients also undergo concurrent radiotherapy 200 cGy/day, 5 days a week for up to 7 weeks (33 fractions), total dose of 6600 cGy.
Period: Overall Study
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Started | 75
Completed | 61
Not Completed | 14
Not completed — Adverse Event | 4
Not completed — Progression | 4
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Three participants did not receive any protocol treatment and were excluded from all analyses.
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 68 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 53
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 12 Months
Description: Percentage of participants who were alive at 12 months.
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Number analyzed (Participants) | 75
percentage of participants | 57 [47 to 70]

2. Secondary Outcome: Response Rate
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
  Response rate is reported as the percentage of participants who achieved each response.
Time Frame: Duration of study (up to 2 years)
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Number analyzed (Participants) | 75
percentage of participants
  Complete Response (CR) | 8
  Partial Response (PR) | 59
  Stable Disease (SD) | 27
  Progressive Disease (PD) | 7

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from registration to disease progression or death of any cause, which ever comes first. The median PFS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Duration of study (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Number analyzed (Participants) | 75
months | 11 [9 to 16]

ADVERSE EVENTS:
Arm/Group | Paclitaxel + Carboplatin + Radiation + Erlotinib
Serious Adverse Events (participants affected / at risk) | 19/75
Other Adverse Events (participants affected / at risk) | 71/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin + Radiation + Erlotinib (N=75)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 14 (15)
Hemolysis (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 3 (4)
Cardiac pain (Cardiac disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 6 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 5 (5)
Ileal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (13)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 1 (2)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 15 (20)
Fever (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (3)
Opportunistic infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 7 (7)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 12 (12)
Lymphocyte count decreased (Investigations) | 8 (8)
Neutrophil count decreased (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 11 (12)
Weight loss (Investigations) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 11 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 13 (14)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (8)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 8 (8)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (4)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (4)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 4 (4)
Personality change (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (20)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (10)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin + Radiation + Erlotinib (N=75)
Hemoglobin decreased (Blood and lymphatic system disorders) | 48 (98)
Hemolysis (Blood and lymphatic system disorders) | 2 (3)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Ear pain (Ear and labyrinth disorders) | 2 (3)
External ear pain (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (3)
Cushingoid (Endocrine disorders) | 1 (2)
Cataract (Eye disorders) | 1 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (3)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 1 (3)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Constipation (Gastrointestinal disorders) | 20 (28)
Diarrhea (Gastrointestinal disorders) | 27 (40)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 12 (13)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 13 (13)
Esophageal pain (Gastrointestinal disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 16 (16)
Fecal incontinence (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (3)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 36 (52)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (25)
Chest pain (General disorders) | 3 (5)
Chills (General disorders) | 3 (3)
Edema limbs (General disorders) | 7 (8)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 65 (126)
Fever (General disorders) | 5 (5)
Gait abnormal (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Pain (General disorders) | 5 (6)
Visceral edema (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 9 (9)
Alkaline phosphatase (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 12 (17)
Blood bilirubin increased (Investigations) | 5 (5)
Creatinine increased (Investigations) | 8 (12)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 28 (43)
Lymphocyte count decreased (Investigations) | 25 (34)
Neutrophil count decreased (Investigations) | 32 (48)
Platelet count decreased (Investigations) | 26 (44)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 17 (21)
Anorexia (Metabolism and nutrition disorders) | 18 (31)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 33 (44)
Dehydration (Metabolism and nutrition disorders) | 10 (12)
Serum albumin decreased (Metabolism and nutrition disorders) | 18 (29)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (10)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 9 (9)
Serum magnesium decreased (Metabolism and nutrition disorders) | 8 (11)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 15 (18)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 17 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (10)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (18)
Dysgeusia (Nervous system disorders) | 8 (11)
Extrapyramidal disorder (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 7 (14)
Peripheral motor neuropathy (Nervous system disorders) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (34)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 6 (11)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 7 (10)
Euphoria (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 12 (17)
Bladder pain (Renal and urinary disorders) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (44)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 48 (88)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (36)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 34 (38)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 2 (4)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (5)
Hypertension (Vascular disorders) | 3 (5)
Hypotension (Vascular disorders) | 3 (4)
Vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less